CLINICAL TRIAL: NCT04805593
Title: Clinical Investigation of the WaveLight® EX500 Excimer Laser for Hyperopic LASIK
Brief Title: Clinical Investigation of the WaveLight® EX500 Excimer Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RFD530-P001
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Hyperopia; Hyperopic Astigmatism
Keywords: LASIK; Refractive errors
MeSH Terms: conditions — Hyperopia; Astigmatism; Refractive Errors | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- WaveLight EX500 excimer laser system (Experimental): Laser-assisted in situ keratomileusis (LASIK) surgery using the WaveLight EX500 excimer laser system
  Interventions: Device: WaveLight EX500 excimer laser system; Procedure: LASIK

INTERVENTIONS:
Device: WaveLight EX500 excimer laser system — FDA approved stationary scanning-spot excimer laser system used during refractive surgery for the treatment of myopia, myopic astigmatism, hyperopia, hyperopic astigmatism, and mixed astigmatism. For this clinical study, the Wavefront Optimized (WFO) Ablation profile of the WaveLight EX500 excimer laser system will be used for bilateral LASIK treatment of hyperopia with and without astigmatism.
Procedure: LASIK — Procedure that reshapes the front part of the eye (cornea) so that light traveling through it is properly focused on the back part of the eye (retina). The procedure will be performed using the WaveLight EX500 excimer laser system.

SUMMARY:
The purpose of this study is to collect efficacy and safety data on the WaveLight EX500 excimer laser system for the correction of hyperopia with and without astigmatism by laser in situ keratomileusis (LASIK) treatment.

DETAILED DESCRIPTION:
Qualified subjects will receive LASIK treatment in both eyes and be followed for 1 year. Subjects will be asked to attend a total of 9 visits (Screening, Surgery, Day 1, Week 1, Month 1, Month 3, Month 6, Month 9, and Month 12). Total expected duration of subject participation is approximately 1 year.

ELIGIBILITY:
Key Inclusion Criteria:

* Intended to treat bilaterally;
* Hyperopia with or without astigmatism as specified in the protocol;
* Stable vision as specified in the protocol;
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Glaucoma;
* Cataracts;
* Previous eye surgery;
* Intent to have monovision treatment;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, Surgical, Study Director — Alcon Research, LLC
Locations (5):
- United States (5):
  - Durrie Vision, Overland Park, Kansas
  - Moyes Eye Center, Kansas City, Missouri
  - Physicians Protocol, Greensboro, North Carolina
  - Vance Thompson Vision ND, West Fargo, North Dakota
  - Mann Eye Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 5 investigative sites located in 1 country (US).
Pre-assignment Details: Of the 44 enrolled, 14 participants were discontinued as screen failures prior to attempted surgery. This reporting group includes all enrolled participants/eyes with attempted surgery (30/60, respectively).
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | WaveLight EX500 Excimer Laser System
Started | 30; 60 eyes
Completed | 30; 60 eyes
Not Completed | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All eyes for which a refractive surgery was attempted with test device (regardless of success or failure).
Arm/Group | WaveLight EX500 Excimer Laser System
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (10.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 29
  Black or African American | 1
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Multi-Racial | 0
  Other | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 26
  Not Reported | 0
  Unknown | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Manifest Refraction Spherical Equivalent (MRSE) Within ±0.50 Diopter (D) at Refractive Stability
Description: A manifest refraction (manual refraction) was performed using a phoropter. The spherical equivalent was calculated by adding the sum of the sphere power with half of the cylinder power. Refractive stability was defined as the latter of two postoperative manifest refractions performed at least 3 months apart (or at 3 months after surgery when compared with the 1-month visit) that meets all the protocol-specified stability requirements. For this endpoint, change in MRSE by less than or equal to 0.50 D was reported. Both eyes contributed data to this analysis.
Time Frame: Up to Month 12 postoperative (Month 1 to Month 3, Month 3 to Month 6, Month 6 to Month 9, and Month 9 to Month 12)
Population: Full Analysis Set (FAS) included all eyes with successful refractive surgery having at least 1 postoperative visit.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | WaveLight EX500 Excimer Laser System
Number analyzed (Participants) | 30
Number analyzed (eyes) | 60
percentage of eyes | 98.3
Statistical Analysis 1: Comparison: WaveLight EX500 Excimer Laser System; Test type: Superiority — Superiority testing was conducted to confirm the proportion is higher than the targeted value of 50%; p < 0.0001, Exact Test of Binomial Proportion

2. Primary Outcome: Percentage of Eyes With MRSE Within ±1.00 D at Refractive Stability
Description: A manifest refraction (manual refraction) was performed using a phoropter. The spherical equivalent was calculated by adding the sum of the sphere power with half of the cylinder power. Refractive stability was defined as the latter of two postoperative manifest refractions performed at least 3 months apart (or at 3 months after surgery when compared with the 1-month visit) that meets all the protocol-specified stability requirements. For this endpoint, change in MRSE by less than or equal to 1.00 D was reported. Both eyes contributed data to this analysis.
Time Frame: Up to Month 12 postoperative (Month 1 to Month 3, Month 3 to Month 6, Month 6 to Month 9, and Month 9 to Month 12)
Population: Full Analysis Set (FAS) included all eyes with successful refractive surgery having at least 1 postoperative visit.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | WaveLight EX500 Excimer Laser System
Number analyzed (Participants) | 30
Number analyzed (eyes) | 60
percentage of eyes | 100.0
Statistical Analysis 1: Comparison: WaveLight EX500 Excimer Laser System; Test type: Superiority — Superiority testing was conducted to confirm the proportion is higher than the targeted value of 75%; p < 0.0001, Exact Test of Binomial Proportion

3. Primary Outcome: Percentage of Eyes Experiencing Ocular Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device (test product). Ocular adverse events were collected for this outcome measure. No hypothesis testing was prespecified for this endpoint.
Time Frame: Up to Month 12 postoperative
Population: Safety Analysis Set: all eyes for which refractive surgery was attempted with the test device (regardless of success or failure).
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | WaveLight EX500 Excimer Laser System
Number analyzed (Participants) | 30
Number analyzed (eyes) | 60
percentage of eyes
  Diplopia | 11.7
  Photophobia | 6.7
  Visual acuity reduced | 3.3
  Ocular hyperaemia | 1.7

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from time of consent to study exit, up to approximately 1 year.
Description: AEs were obtained through solicited and spontaneous comments from the subjects and through observations by the investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all subjects/eyes.
Groups:
- Pretreament: AEs in this group occurred prior to treatment with the WaveLight EX500 excimer laser system.
- WaveLight EX500 Excimer Laser System - Ocular: AEs in this group occurred after attempted treatment with the WaveLight EX500 excimer laser system and include ocular events in the study eye.
- WaveLight EX500 Excimer Laser System - Systemic: AEs in this group occurred after attempted treatment with the WaveLight EX500 excimer laser system and include overall systemic events.
Arm/Group | Pretreament | WaveLight EX500 Excimer Laser System - Ocular | WaveLight EX500 Excimer Laser System - Systemic
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/60 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 2/60 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 10/60 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreament (N=30) | WaveLight EX500 Excimer Laser System - Ocular (N=60) | WaveLight EX500 Excimer Laser System - Systemic (N=30)
Visual acuity reduced (Eye disorders) | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreament (N=30) | WaveLight EX500 Excimer Laser System - Ocular (N=60) | WaveLight EX500 Excimer Laser System - Systemic (N=30)
Diplopia (Eye disorders) | 0 | 7 | 0
Photophobia (Eye disorders) | 0 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to study.

DOCUMENTS (2):
  • Study Protocol (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/93/NCT04805593/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/93/NCT04805593/SAP_001.pdf